CLINICAL TRIAL: NCT07157332
Title: Dysregulation of Iron Metabolism in Obese Individuals and Its Implications for Metabolic Health
Brief Title: Iron Metabolism in Obesity
Acronym: IRON-XL
Status: Not yet recruiting | Type: Observational
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: Fundación Santos y de la Garza Evia, IBP (Unknown)
Responsible Party: Sponsor
Other Study IDs: IPI-D
Record Dates: First submitted 2025-08-07; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity (Disorder)
Keywords: Obesity; Weight loss; Iron metabolism; Metabolic health; Bariatric surgery; Body composition; Inflammation markers; Dietary assessment
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens collected and retained in this study include: whole blood samples for serum and plasma separation, used for biochemical, hematological, and immunological analyses; subcutaneous and visceral adipose tissue biopsies obtained perioperatively for assessment of cellular iron metabolism and oxidative stress; stool samples for gut microbiota metagenomic sequencing; and urine samples for pregnancy testing prior to DEXA scans. Blood samples will be aliquoted and stored at -80ºC for future analyses. Tissue and stool samples will be processed according to standardized protocols to preserve DNA integrity and cellular components.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iron Deficiency Group: Participants with obesity who meet the World Health Organization criteria for systemic iron deficiency, defined as serum ferritin < 15 µg/L or < 70 µg/L in presence of inflammation, and/or elevated transferrin receptor levels (>8.2 µg/L). These participants undergo bariatric surgery and are followed prospectively for changes in iron metabolism, oxidative stress, inflammation, and metabolic health.
  Interventions: Procedure: Bariatric Sleeve Surgery
- Non-Iron Deficiency Group: Participants with obesity without systemic iron deficiency according to WHO standards, with normal serum ferritin and transferrin receptor levels. They undergo bariatric surgery and are followed in parallel to the iron deficiency group to compare outcomes in iron metabolism, oxidative stress, inflammation, and metabolic health over 6 months post-surgery.
  Interventions: Procedure: Bariatric Sleeve Surgery

INTERVENTIONS:
Procedure: Bariatric Sleeve Surgery — Participants undergo a restrictive bariatric procedure called sleeve gastrectomy, performed by experienced surgeons. This procedure involves surgical reduction of the stomach size to aid in weight loss. The study observes outcomes related to iron metabolism, body composition, and biochemical markers over six months post-surgery. No additional interventions or treatments are applied as part of the study protocol; the surgery is part of routine clinical care.
  Other Names: Sleeve Gastrectomy

SUMMARY:
This study consists of two phases and aims to understand how obesity and systemic iron deficiency affect iron accumulation in important organs such as the liver and heart, as well as oxidative stress in fat tissue cells. In Phase 1, researchers will compare individuals with obesity who have iron deficiency to those without, to see if there are differences in the amount of iron stored in the liver and heart, measured by magnetic resonance imaging (MRI), and in oxidative stress and labile iron in visceral and subcutaneous fat tissue, assessed through biopsies. Phase 2 is a six-month prospective cohort study following the same individuals after they undergo bariatric surgery, a weight-loss surgery. The goal is to evaluate whether weight and fat loss normalize iron accumulation in the liver and heart, reduce oxidative stress, improve systemic iron metabolism, enhance blood sugar control, support liver function, modulate chronic inflammation, and restore gut microbiota diversity. Researchers will compare these health changes between individuals with and without iron deficiency. The study includes adults aged 18 to 50 with obesity living in the metropolitan area of Monterrey, Mexico, who are scheduled for laparoscopic sleeve gastrectomy surgery and agree to participate. The findings could improve understanding of how iron metabolism interacts with obesity-related complications and may lead to better treatments and management strategies for people with obesity and iron deficiency.

DETAILED DESCRIPTION:
This is a prospective observational cohort study designed to evaluate changes in clinical, biochemical, and dietary variables related to iron status in adult individuals undergoing restrictive bariatric surgery (laparoscopic sleeve gastrectomy or adjustable gastric banding) in the urban area of Monterrey, Mexico. The main objective is to assess whether iron status prior to surgery influences weight loss success, inflammatory response, and overall health-related quality of life in the six months following surgery.

A total of 50 participants (25 with iron deficiency and 25 without, defined according to WHO standards) will be enrolled. Participants will be classified into groups based on baseline iron status measured using routine preoperative laboratory data. Eligibility criteria include age between 18 and 50 years, premenopausal women, BMI between 35 and 45 kg/m², and eligibility for restrictive bariatric surgery according to international guidelines. Exclusion criteria include prior bariatric surgery, severe anemia (Hb < 100 g/L), medical conditions that may affect inflammation or iron metabolism, chronic liver disease, recent pregnancy or lactation, recent significant weight loss (>10% in the last 6 months), shift work, and high levels of physical activity (>10 hours/week).

All participants will be followed for 6 months after surgery. Outcome assessments include anthropometric measurements, laboratory parameters (hemoglobin, ferritin, CRP, among others), dietary intake, and patient-reported outcomes. Dietary intake will be assessed using MyFitnessPal, a mobile app for dietary tracking, with standardized food entries labeled "IRONXL" based on the Mexican food composition database. Participants will be trained to enter food items accurately and consistently. Data from MyFitnessPal will be exported to obtain nutrient intake data.

Quality of life and general health status will be measured using the PROMIS Global Health questionnaire, a validated 10-item tool. A structured case report form will collect demographic, medical history, and lifestyle data. Blood samples will be collected and stored for potential future research purposes, pending optional consent by participants.

The study will be conducted at the Zambrano Hellion Medical Center, TecSalud. The research team includes qualified surgeons and investigators trained in Good Clinical Practice (GCP). Data quality assurance procedures will include double-entry verification of questionnaire data, standardized anthropometric assessments, and laboratory analyses conducted in accredited clinical laboratories. A Manual of Procedures (MOP) guides all data collection processes.

Missing data will be managed through multiple imputation when appropriate, and all analyses will be conducted according to a pre-specified Statistical Analysis Plan (SAP). The primary outcome is change in weight (kg and % of initial body weight) over 6 months. Secondary outcomes include change in hemoglobin, ferritin, CRP, dietary iron intake, and PROMIS scores.

The sampling method is non-probabilistic and based on convenience sampling of patients scheduled for surgery who meet the eligibility criteria and agree to participate voluntarily. All participants will provide written informed consent before any study procedures.

Optional consent will be obtained for the long-term storage and future analysis of biospecimens (whole blood, serum). These samples may be used in future research related to iron metabolism, inflammation, and nutrition. Participants who decline this optional component will still be eligible to participate in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 50 years.
* Premenopausal women (defined as no absence of menstruation in the past 12 months).
* Body Mass Index (BMI) between 35 and 45 kg/m² at recruitment.
* Scheduled to undergo bariatric surgery via sleeve gastrectomy or laparoscopic adjustable gastric banding (LAGB), with indications aligned with international guidelines. Bariatric surgery eligibility includes:

  1. BMI between 35 and 45 kg/m² with the presence of obesity-related comorbidities (medical, physical, or psychosocial conditions), and a history of unsuccessful attempts at sustained weight loss through non-surgical means.
  2. Adequately informed, understanding and accepting the potential risks and benefits of the procedure, and expressing commitment to adhere to long-term dietary and physical activity recommendations post-surgery.
* Willing to maintain consistent dietary iron intake and refrain from taking any iron supplements other than those prescribed by the attending surgeon throughout the study duration.
* Not pregnant during the study period or in the six months prior to enrollment, and not planning to become pregnant for at least 3 months after the final study visit (at 6 months).
* Not breastfeeding in the six weeks prior to enrollment, nor planning to breastfeed during the study.
* No significant weight loss (≥10% of body weight) in the six months prior to the pre-surgical evaluation.
* Signed informed consent.
* No night shift work during the two weeks prior to the baseline visit or at any point during the study (night shift defined as work performed between 12:00 AM and 6:00 AM).
* Not engaging in strenuous physical activity ≥10 hours per week.

Exclusion Criteria:

* Participants who have undergone any bariatric procedure other than LAGB or sleeve gastrectomy.
* Severe anemia (defined as hemoglobin <100 g/L).
* History of previous surgical obesity treatments.
* Presence of significant medical conditions that may affect iron status or inflammatory markers independently of obesity, including but not limited to: cancer, HIV/AIDS, inflammatory bowel disease, gastrointestinal bleeding, rheumatoid arthritis, and chronic kidney disease (per investigator's judgment).
* Diagnosed abnormalities in iron metabolism based on routine pre-surgical blood samples and unrelated to obesity (e.g., thalassemia).
* History of frequent blood transfusions.
* Chronic liver disease (e.g., alcoholic liver disease, hepatitis C-related liver disease).
* Use of medications that could interfere with study measurements (per investigator's judgment).
* Women consuming ≥14 alcoholic beverages per typical week or men consuming >21 alcoholic beverages per typical week.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of obese adults scheduled for restrictive sleeve bariatric surgery residing in the urban area of Monterrey, Mexico, who voluntarily agree to participate in the study over a 6-month follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Body Weight Loss at 6 Months Post-Surgery | Measured at baseline (pre-surgery) and 6 months post-surgery.
  Proportion of initial body weight lost by each participant, calculated as ((initial weight - weight at 6 months) / initial weight) × 100. This measure is used to assess the effectiveness of bariatric sleeve surgery and to evaluate differences between participants with and without iron deficiency.

SECONDARY OUTCOMES:
Percentage of total body fat | Baseline, 3 months, and 6 months after baseline visit.
  Measurement of total body fat percentage using Dual-Energy X-ray Absorptiometry (DEXA) scans.
Lean mass | Baseline, 3 months, and 6 months after baseline visit.
  Measurement of total lean body mass in kilograms using DEXA scans.
Bone mineral density | Baseline, 3 months, and 6 months after baseline visit.
  Measurement of bone mineral density using DEXA scans.
Changes in gut microbiota composition | Baseline and 6 months after baseline visit.
  Analysis of fecal samples by 16S rDNA sequencing to evaluate changes in gut microbiota diversity and composition at baseline and 6 months post-surgery.
Blood pressure | At baseline, 1 month, 3 months, and 6 months post-baseline.
  Measurement of blood pressure using an automated monitor.
Resting heart rate | Baseline, 1 month, 3 months, and 6 months post-baseline.
  Measurement of resting heart rate using an automated monitor.
Fasting plasma glucose | Baseline, 3 months, and 6 months post-baseline.
  Measurement of fasting plasma glucose concentration from venous blood samples.
Insulin | Baseline, 3 months, and 6 months post-baseline.
  Measurement of fasting plasma insulin concentration from venous blood samples.
Total cholesterol | Baseline, 3 months, and 6 months post-baseline.
  Measurement of total cholesterol
LDL cholesterol | Baseline, 3 months, and 6 months post-baseline.
  Measurement of LDL cholesterol
HDL cholesterol | Baseline, 3 months, and 6 months post-baseline.
  Measurement of HDL cholesterol
Triglycerides | Baseline, 3 months, and 6 months post-baseline.
  Measurement of triglycerides
HOMA-IR index | Baseline, 3 months, and 6 months post-baseline.
  Calculation of insulin resistance using fasting plasma glucose and insulin values.
C-reactive protein | Baseline, 3 months, and 6 months post-baseline.
  Measurement of serum C-reactive protein concentration using high-sensitivity assay.
TNF-α | Baseline, 3 months, and 6 months post-baseline.
  Measurement of TNF-α
IL-6 | Baseline, 3 months, and 6 months post-baseline.
  Measurement of IL-6
IL-1β | Measurement of TNF-α, IL-6, and IL-1β
  Measurement of IL-1β
Leptin | Baseline, 3 months, and 6 months post-baseline.
  Measurement of leptin

OTHER OUTCOMES:
Quality of life evaluation using the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health 10-item questionnaire | Baseline and 6 months post-baseline.
  Assessment of general health, mental health, fatigue, pain, and functionality using the PROMIS Global Health 10-item questionnaire. Each item is scored on a 1-5 Likert scale, with higher scores indicating better health status. Raw scores are converted to standardized T-scores, which range from 0 to 100. For all domains, higher scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Cepeda Lopez, PhD, Principal Investigator — Fundación Santos y de la Garza Evia, IBP
Locations (1):
- Fundación Santos y de la Garza Evia, IBP, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications arising from this study, including data on clinical, anthropometric, and laboratory outcomes, will be shared after de-identification
Supporting Information: Study Protocol, SAP, Analytic Code